CLINICAL TRIAL: NCT05422274
Title: Evaluating the Efficacy and Safety of Transcranial Pulse Stimulation on Young Adolescents with Attention-Deficit-Hyperactivity Disorder- a Pilot Randomized, Double-blinded, Sham-controlled Trial
Brief Title: Effect of Transcranial Pulse Stimulation on ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HongKongPU_HSEARS20220518006
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-09

CONDITIONS: ADHD
Keywords: Efficacy and Safety; Transcranial Pulse Stimulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, sham-controlled trial.
Who Masked: Participant, Investigator
Masking Description: Double-blind. Participants and interventionists will be blinded to the random allocation to either the verum TPS group or the sham TPS group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Pulse Stimulation (TPS group) (Experimental): Subjects in the TPS group will be given 6 verum TPS sessions (Pulse: 800 / session) across two weeks time, with 3 sessions per week.
  Interventions: Device: Transcranial Pulse Stimulation
- Sham TPS Group (Sham Comparator): Subjects in the Sham TPS group will be given 6 sham TPS sessions across two weeks time, with 3 sessions per week.
  Interventions: Device: Transcranial Pulse Stimulation

INTERVENTIONS:
Device: Transcranial Pulse Stimulation — A total of 36 participants (both TPS group and the sham-control group) will receive six 30 minute-TPS sessions (800 pulse in each session, total: 4800 pulse) in 2 weeks' time (i.e., 3 sessions (Monday, Wednesday, Friday) per week, total: 3 hours), on a 1: 1 allocation ratio. Participants will be followed up immediately after the post-stimulation and at 1-month and 3-month period after the intervention. A 2-week TPS intervention alongside with 3-month follow-up is sufficient enough to test the effects of TPS on improving inattention and hyperactivity .

SUMMARY:
This is the first nationwide study using Transcranial Pulse Stimulation to evaluate its efficacy and safety on 30 young adolescents with ADHD. Six verum/ shamTPS sessions will be delivered to all subjects on a 1: 1 ratio, balanced by gender and age. Attention deficit, hyperactivity, impulsivity, and oppositional defiance will be the primary outcome. Secondary outcomes include ADHD severity, frequency of inattention, hyperactivity, impulsivity, executive function and neural connectivity changes via neuroimaging. Results emerging from this study will generate new knowledge to ascertain whether TPS can be used as a top-on treatment in ADHD.

DETAILED DESCRIPTION:
Objectives of the study

1. To evaluate the efficacy and safety of TPS on young adolescents (12-17 years) with ADHD in Hong Kong.
2. To examine the association between TPS and ADHD core symptom severity, executive function, inattention, hyperactivity, impulsivity, and oppositional defiance.
3. To examine the brain functional connectivity changes immediately after the 2-week TPS treatment via neuroimaging.

Expected outcomes/Hypotheses:

1. Participants in the verum TPS group or the sham TPS group will have <5% somatic discomfort in the 2-week TPS intervention and that TPS is a safe intervention on young adolescents with ADHD.
2. Participants in the verum TPS group will have 30% reduction in the Swanson, Nolan, and Pelham Rating Scale (SNAP IV score) (i.e., attention deficit, hyperactivity impulse and oppositional defiance) after 2-weeks TPS treatment compared with the sham TPS group and be maintained at the 1- month & 3-month follow-up.
3. Participants in the verum TPS group will have 30% improvement in the ADHD symptoms and behaviour compared with the sham TPS group after 2-weeks TPS treatment and be maintained at the 1-month & 3-month follow-up.
4. Participants in the verum TPS group will have 30% improvement in executive function after 2 weeks TPS treatment compared with the sham TPS group and be maintained at the 1-month & 3-month follow-up.
5. Participants in the verum TPS group will have 30% improvement in both attention deficit & reduction in hyperactivity, impulsivity after 2 weeks TPS treatment compared with the sham TPS group, and be maintained at the 1 month & 3-month follow-up.
6. Participants in the verum TPS group will have more brain connectivity changes after 2-weeks TPS compared with the sham TPS group and be maintained at the 1 month & 3-month follow-up.

Design: This is a two-armed, randomized, double-blind, sham-controlled trial.

Sample size:

To the best of our knowledge, there is no interventional study evaluating the efficacy of TPS on ADHD. Based on our previous open label pilot RCT 37 evaluating TPS on adults with Major Depressive Disorder that showed a large effect size (f = 0.47), we hypothesize a large effect of TPS in this study. We used G*power version 3.1.9.4 to calculate the target sample size. With a statistical power of 95% and a statistical significance level at 0.05 to detect a large between-groups effect size (f) of 0.47 with 4 measurement time points, each group will require 15 subjects. A total sample of 30 is required in this trial. The attrition rate in our pilot MDD trial was 0%. We expect that the attrition rate in this ADHD trial would be <5%. Subject dropping out the 2-week intervention period will be replaced by another enrolled subject in this pilot study.

Intervention (Transcranial Pulse Stimulation) Purpose of the intervention: The key tenets of the TPS intervention is neuromodulation, i.e., using ultrasound-based brain stimulation techniques to modulate the human brain in a focal and targeted manner. Intervention dose: Each participant should have the pre-treatment MRI scan performed in the University Research Facility in Behavioural and Systems Neuroscience, PolyU prior coming to the first intervention session. All participants (both TPS group and the sham-control group) will receive six 30 minute-TPS sessions (800 pulse in each session, total: 4800 pulse) in 2 weeks' time. Participants will be followed up immediately after post-stimulation in Week 2, and at 1-month and 3- month period after the intervention. The investigators believe that a 2-week TPS intervention is sufficient enough to test the effects of TPS on improving inattention and hyperactivity.

ELIGIBILITY:
Inclusion Criteria:

1. have a confirmed diagnosis of ADHD according to the 5th edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-5) of the American Psychiatric Association;
2. ethic Chinese, aged 12-17, with no co-morbidity of other mental disorders (e.g., Intellectual Disability Disorder) and organic brain diseases that affected cognitive functions;
3. no severe systemic diseases including heart, liver, lung, and kidney diseases;
4. have an IQ >80 by Stanford-Binet Intelligence Scales, 5th Edition (SB-5);
5. written consent by parents.

Exclusion Criteria:

1. SNAP IV score <1;
2. not taking ADHD medications in the past 2-4 weeks;
3. treated with TMS/rTMS/tDCS or electroconvulsive therapy in the past 12 months;
4. taking monoamine oxidase inhibitors in the past 14 days;
5. have a history of epilepsy, brain trauma, brain surgery/brain tumour, brain aneurysm or other concomitant unstable major medical conditions like haemophilia or other blood clotting disorders or thrombosis;
6. significant communicative impairments;
7. having metal implants in the brain treatment region /artificial cardiac pacemaker in-situ;
8. taking corticosteroid treatment within the last six weeks before the first TPS treatment;
9. have a history of micro-cavernomas.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Attention deficit, hyperactivity impulse and oppositional defiance | Changes in SNAP-IV scores from baseline at 3 months
  The Swanson, Nolan, and Pelham Rating Scale (SNAP IV) will be used to measure participants' attention deficit, hyperactivity impulse and oppositional defiance. SNAP IV consists of 26 items summarized into three factors: attention deficit, hyperactivity impulse, and oppositional defiance. Parents based on their general impressions on their children and rate the severity of symptoms on a Likert scale (0-3). Mean score <1 indicate "normal" or "remission"; Mean score of 1 is defined as the demarcation for attention deficit and hyperactivity impulsivity; mean score >2 indicated "abnormal".
  SNAP-IV is a reliable and valid scale used in RCTs and has good psychometric properties in the Chinese population.

SECONDARY OUTCOMES:
Clinical global impression | Changes in CGI from baseline at 3 months
  CGI-S is a 7-point clinician rating scale is based upon observed and reported symptoms, behaviour, and function in the past seven days. CGI-I is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Executive function | Changes in Stroop test from baseline at 3 months
  Stroop test is a neuropsychological test commonly used to assess the inhibition control component of executive function and test the subject's ability to inhibit cognitive interference that occurs when the processing the target stimulus feature is impeded by the simultaneous processing of a second stimulus attribute.
The ADHD Rating Scale-IV | Changes in ADHD RS-IV from baseline at 3 months
  ADHD RS-IV is a widely used ADHD scale comprising 18 items. Participant's parent rates the frequency of each symptom on the scale. Each item scores on a 4-point Likert scale of 0-3 (0: never or rarely; 1: sometimes; 2: often; 3: very often). The 9 odd items evaluate attention deficits, composing the Inattention subscale (or IA); the 9 even items evaluate Hyperactivity Impulsivity, composing the Hyperactivity Impulsivity (or HI) subscale; the total score is the sum of all the scores on the 18 items. The ADHD RS-IV is a reliable and valid scale in the Chinese population.
Neuroimaging | MRI will be assessed at baseline at immediately and 2 weeks after post-stimulation
  Participants will receive pre and post treatment MRI scan to measure any changes in structural and functional connectivity changes in the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Teris Cheung, PhD, Principal Investigator — HongKongPolyU
Locations (1):
- School of Nursing HongKongPolyU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheung T, Yee BK, Chau B, Lam JYT, Fong KH, Lo H, Li TMH, Li AM, Sun L, Beisteiner R, Cheng CPW. Efficacy and safety of transcranial pulse stimulation in young adolescents with attention-deficit/hyperactivity disorder: a pilot, randomized, double-blind, sham-controlled trial. Front Neurol. 2024 May 9;15:1364270. doi: 10.3389/fneur.2024.1364270. eCollection 2024. PMID 38784916
- [Derived] Cheung T, Chau B, Fong KH, Lam JYT, Lo H, Li MH, Li AMMC, Beisteiner R, Lei S, Yee BK, Cheng CPW. Evaluating the efficacy and safety of transcranial pulse stimulation on adolescents with attention deficit hyperactivity disorder: Study protocol of a pilot randomized, double-blind, sham-controlled trial. Front Neurol. 2023 Mar 28;14:1076086. doi: 10.3389/fneur.2023.1076086. eCollection 2023. PMID 37056363